CLINICAL TRIAL: NCT04878081
Title: The Relationship Between Day and Night Hot Flash During Menopause and Different Traditional Chinese Constitution Types in Women
Brief Title: Day and Night Hot Flash During Menopause
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH109-REC1-184
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Menopause

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: hot flush — Hot Flash Diaries to record the change of daily hot flush symptoms for 30 days. The Hot Flash Related Daily Interference Scale to record how much did hot flush effect daily life.
  The Kupperman menopausal index to evaluate the severity of menopausal symptoms. The Pittsburgh Sleep Quality Index to evaluate sleep disorder. Wireless temperature monitor to record hot flush and body temperature during sleeping.
  Classify patients' traditional Chinese constitution by using Physical classification and judgment self-test table.

SUMMARY:
We use Hot Flash Diaries to record the change of daily hot flush symptoms, The Hot Flash Related Daily Interference Scale to record how much did hot flush effect daily life, the Kupperman menopausal index to evaluate the severity of menopausal symptoms, the Pittsburgh Sleep Quality Index to evaluate sleep disorder, wireless temperature monitor to record hot flush and body temperature during sleeping, and classify patients' traditional Chinese constitution by using Physical classification and judgment self-test table. With these evaluations, we can take apart of different syndromes with different symptom of menopause, thus to confirm the specificity and the severity of menopausal hot flush, and give patients correct treatment.

DETAILED DESCRIPTION:
Menopause syndrome or Climacteric syndrome is defined as decreasing function of ovarian follicles during menopause. This situation leads to the decreased concentration of estrogen, and causes a series of physical and psychological symptoms, with main symptoms of hot flush, night sweats, dizziness or headache, limbs soreness, insomnia, anxiety and depression. Approximately 40-60 % of menopausal women have the problem of menopausal symptoms, these symptoms severely affect the life quality of post-menopausal women. We use Hot Flash Diaries to record the change of daily hot flush symptoms, The Hot Flash Related Daily Interference Scale to record how much did hot flush effect daily life, the Kupperman menopausal index to evaluate the severity of menopausal symptoms, the Pittsburgh Sleep Quality Index to evaluate sleep disorder, wireless temperature monitor to record hot flush and body temperature during sleeping, and classify patients' traditional Chinese constitution by using Physical classification and judgment self-test table. With these evaluations, we can take apart of different syndromes with different symptom of menopause, thus to confirm the specificity and the severity of menopausal hot flush, and give patients correct treatment.

ELIGIBILITY:
Inclusion Criteria:

* not accept Chinese medicine therapy for last 3 months
* 40-55 years old female
* prolonged menstruation with hot flush, night sweats or insomnia
* regular night sleep habit
* not take oral contraceptive pill for last 6 months
* no smoking, alcohol, drug abused

Exclusion Criteria:

* any types of Systemic disease
* any chronic disease under medicine control
* any mental disorder
* pregnant women

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: menopausal women
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
the change of daily hot flush symptoms | 30 days
  the change of daily hot flush symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Yu Su, M.D. Ph.D., Study Director — 886-4-22052121 Ext. 4561
Locations (1):
- CMUH, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided